CLINICAL TRIAL: NCT02308475
Title: Myocardial Stress Perfusion Computed Tomography in the Evaluation of Patients With Acute Chest Pain Using a Novel 3rd Generation Dual-source CT System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New study with a similar endpoint/protocol was developed (see NCT03103061).
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, U. Joseph Schoepf, MD, Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro31584
Record Dates: First submitted 2014-11-21; First posted 2014-12-04 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myocardial Stress CT Perfusion (Experimental): Dynamic volume CT myocardial perfusion using the experimental scanner (Force, Siemens), applying the "dynamic shuttle" mode will be used to rapidly cover the entire cardiac anatomy during infusion of a contrast medium bolus for monitoring bolus passage through the left ventricular myocardium.
  Interventions: Device: Somatom Force CT Scanner

INTERVENTIONS:
Device: Somatom Force CT Scanner — Dynamic CT perfusion of the heart

SUMMARY:
To assess the ability of a novel 3rd generation dual-source CT system to demonstrate myocardial perfusion in a cohort of patients presenting to the Chest Pain Center with acute chest pain.

DETAILED DESCRIPTION:
The investigators will assess the latest generation of CT scanner for heart disease detection. On this new machine the investigators will analyse the ability of the machine to show the delivery of blood to the heart muscle. Results will be compared with the results from the gold standard test for myocardial perfusion imaging, which is an imaging test that shows the blood supply to the heart muscle. Further analyses will record the amount of radiation, which is how the CT machine acquires images, and compare the amount of radiation necessary to produce images to previous CT systems. With this new CT system there should be reductions in the amount of radiation dose compared to previous systems.

ELIGIBILITY:
Inclusion Criteria:

* Subject must present with symptoms of acute but atypical or recurrent chest pain.
* Subject must have been referred for cardiac CT angiography OR subject must have undergone clinically indicated SPECT with positive or equivocal findings OR subject must have undergone clinically indicated SPECT with prior cardiac CT angiography that showed moderate or severe stenosis.
* Subject must be 18-85 years of age.
* Subject must provide written informed consent prior to any study-related procedures being conducted.
* Subject must be willing to comply with all clinical study procedures.

Exclusion Criteria:

* Subject is a pregnant or nursing female.
* Subject has severe asthma or COPD requiring frequent inhaler use.
* Subject has prior diagnosis of obstructive CAD that has not been revascularized.
* Subject with implanted rhythm devices (pacemaker, defibrillator).
* Subject has significant arrhythmia.
* Subject has high grade heart block.
* Subject has resting heart rate < 45 bpm, systolic blood pressure <90 mm Hg, or has consumed caffeine within the last 12 hours.
* Subject has an acute psychiatric disorder.
* Subject is unwilling to comply with the requirements of the protocol.
* Subject has previously entered this study.
* Subject has an allergy against iodinated contrast or pharmaceutical stressors used in this study.
* Subject suffers from claustrophobia.
* Subject has impaired renal function (creatinine > 1.5 mg/dl).
* Subject is in unstable condition.
* ST-elevations, new transient ST changes greater than 0.05mV or T-wave inversions with symptoms.
* Subject cannot safely be administered Lexiscan per prescribing information as as determined by investigator.
* Subject has received interventional (PCI, stenting) or surgical (CABG) treatment that may alter the cardiac condition regarding myocardial perfusion status and/or stenosis degree between cardiac CTA, SPECT, and/or CT stress perfusion studies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07-06 (Actual); Study Completion 2015-07-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Myocardial Stress CT Perfusion
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Myocardial Stress CT Perfusion
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 34.5 [33 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2
Height [Mean (Full Range); unit: inches] | 67 [65 to 69]
Weight [Mean (Full Range); unit: lbs] | 248.5 [241 to 256]

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy of Dynamic Perfusion CT
Description: The diagnostic accuracy of dynamic perfusion CT of the heart for evaluation of perfusion, viability and function during stress and rest will be compared with SPECT myocardial perfusion imaging using p-values for comparison of reader specific values, calculated by means of the McNemar test.
Time Frame: 1 Day
Population: The planned statistical analyses were not performed.
Arm/Group | Myocardial Stress CT Perfusion
Number analyzed (Participants) | 0

2. Secondary Outcome: CTMP/SPECT MPI Disagreement
Description: Evaluate the accuracy of CT myocardial perfusion and SPECT using a stress/rest and delayed enhancement MRI examination as gold-standard by means of Kappa analysis
Time Frame: 1 Day
Population: The planned statistical analyses were not performed.
Arm/Group | Myocardial Stress CT Perfusion
Number analyzed (Participants) | 0

3. Secondary Outcome: Radiation Dose
Description: Assess the radiation dose (in mGy) delivered with the myocardial perfusion CT comparing the results with those obtained at SPECT.
Time Frame: 1 Day
Population: The planned statistical analyses were not performed.
Arm/Group | Myocardial Stress CT Perfusion
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Myocardial Stress CT Perfusion
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myocardial Stress CT Perfusion (N=2)
Chest Pain (General disorders) | 1 (1) — ED visit for chest pain radiating to the shoulder and abdomen

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No